CLINICAL TRIAL: NCT04859686
Title: Acupuncture and Meditation for Wellness (AMWELL)
Brief Title: Acupuncture and Mindfulness Based Stress Reduction for Wellness
Acronym: AMWELL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HP-00043308
Record Dates: First submitted 2020-10-23; First posted 2021-04-26 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-04

CONDITIONS: PTSD
Keywords: PTSD; Depression; Acupuncture; Mindfulness-based stress reduction; Child abuse survivors
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Mindfulness-Based Stress Reduction; Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Participants underwent intervention.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction; Procedure: Acupuncture Treatment
- Waitlist (No Intervention): Participants received no intervention.

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The MBSR program included weekly 2.5-hour sessions in a group format over eight weeks, plus a 1-day retreat. Formal practices included several types of meditation, such as mindful breathing, sitting meditation, walking meditation, gentle hatha yoga, body scan, and mindful awareness. Participants were asked to practice at home for 20 minutes daily, six days a week.
  Other Names: MBSR
  Arms: Treatment
Procedure: Acupuncture Treatment — Participants received two treatments per week over eight weeks, 35-40 minutes each.
  At each treatment, participants were treated with 10 body and two ear points: seven major points on either the front or back of the body. The treatment position alternated between sessions, such that the first session was on the back, with the next session on the front, unless a physical limitation prevented alternation.
  Arms: Treatment

SUMMARY:
AMWELL is a randomized, waitlist-controlled, pilot study to evaluate the comparative efficacy of Mindfulness Based Stress Reduction (MBSR) and Acupuncture (AT) to Wait-List Control (WL) in adult female survivors of childhood sexual abuse (CSA) experiencing symptoms of psychological distress.

DETAILED DESCRIPTION:
Female CSA survivors at least 21 years old were recruited from newspaper ads, radio programs, study websites and various public announcements in the Baltimore, Md and surrounding area between September, 2008 to October, 2009.

ELIGIBILITY:
Inclusion Criteria:

* Female survivors of childhood sexual assault reported in a clinical interview (e.g., age at which the abuse began and continued, frequency and duration, and the perpetrator)
* At least 21 years old
* Ability to read and write in English
* Under the care of a licensed psychotherapist or physician for study duration
* Clinical approval for acupuncture or MBSD
* Ability to attend 80% of the sessions
* Willingness to practice skills 20-30 minutes per day, six days a week
* If taking psychotropic medication, on a stable dose for 30 days prior to baseline
* A score of 0.5 or greater on the Brief Symptom Inventory (BSI)

Exclusion Criteria:

* Any major illness or psychiatric disorder
* Symptom severity as evidenced by a CGI-S score of 6 or 7
* Current suicidal ideation
* Active alcoholism or drug dependency
* Current enrollment in another clinical trial
* Major surgery scheduled
* Plans to move from the area during the 12-week study period
* Current pregnancy, plans to become pregnant, or no means of birth control

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2009-10-01 (Actual); Study Completion 2010-10-30 (Actual)

PRIMARY OUTCOMES:
PTSD Checklist 4 (PCL-IV) Score | Week 4, 8 and 12
  PCL-IV is a self-report measure of 17 DSM-IV symptoms of PTSD. A total symptom severity score (range = 17-85) was obtained by summing the scores from each of the 17 items that have response options ranging from 1 "Not at all" to 5 "Extremely. Higher scores indicate worse symptoms of PTSD. Participants were evaluated by a study coordinator at a baseline visit, at 4 weeks for a mid-treatment measure, at 8 weeks for a posttreatment measure, and at 12 weeks for a one month follow-up assessment. Effects of the intervention were assessed using repeated measures, mixed model analysis of mean scores for each of the outcomes at baseline, 4, 8, and 12 weeks. The magnitude of treatment effect was calculated by Cohen's d for each treatment defined as the baseline to 8 week or 12 week change in mean score divided by the standard deviation of the change in scores.
Beck Depression Inventory (BDI-II) Score | Week, 4, 8 and 12
  The 21-item BDI-II is a widely-used, standardized, validated self-reporting measure of depressive symptom severity. It addresses affective, behavioral, biological, cognitive, and motivational symptoms of depression. Participants rated statements from 0 to 3 to indicate the level which best described the severity of the symptoms experienced. The ratings were summed to a total score, with ranges of 4-9 indicating "normal," 10-18 "mild," 9-29 "moderate to severe," and ≥ 30 indicating "severe." Scores range from 0 - 40. Higher scores indicate worse depressive symptoms. Effects of the intervention were assessed using repeated measures, mixed model analysis of mean scores for each of the outcomes at baseline, 4, 8, and 12 weeks. The magnitude of treatment effect was calculated by Cohen's d for each treatment defined as the baseline to 8 week or 12 week change in mean score divided by the standard deviation of the change in scores.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI Score | Week 4, 8 and 12
  The PSQI is a 19-item self-reported inventory providing measures of daytime dysfunction, sleep latency, duration, disturbance, quality, and efficiency, which are arranged into seven component scores. Each item is rated 0 (best) to 3 (worst); the component sums are added together, ranging from 0 (worst) to 21 (best), providing a global PSQI score. Higher scores indicate worse sleep quality.
The Mindfulness Attention Awareness Scale (MAAS) Score | Week 4, 8 and 12
  The 15-item self-report MAAS measures mindfulness as open or receptive awareness and attention to the present. The questions ask about daily experiences (e.g., I snack without being aware that I'm eating.), with answers being measured on a Likert-scale of 1 (almost always) to 6 (almost never). Scores range from 15 - 90. Higher scores reflect higher levels of mindfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Berman, MD, Principal Investigator — University of Maryland, Baltimore

REFERENCES:
- [Background] Afifi TO, Taillieu T, Zamorski MA, Turner S, Cheung K, Sareen J. Association of Child Abuse Exposure With Suicidal Ideation, Suicide Plans, and Suicide Attempts in Military Personnel and the General Population in Canada. JAMA Psychiatry. 2016 Mar;73(3):229-38. doi: 10.1001/jamapsychiatry.2015.2732. PMID 26817953
- [Background] Silver KE, Levant RF. An appraisal of the American Psychological Association's Clinical Practice Guideline for the Treatment of Posttraumatic Stress Disorder. Psychotherapy (Chic). 2019 Sep;56(3):347-358. doi: 10.1037/pst0000230. PMID 31282711
- [Background] Bedard-Gilligan M, Jaeger J, Echiverri-Cohen A, Zoellner LA. Individual differences in trauma disclosure. J Behav Ther Exp Psychiatry. 2012 Jun;43(2):716-23. doi: 10.1016/j.jbtep.2011.10.005. Epub 2011 Oct 29. PMID 22080869
- [Background] Beck, A. T., Steer, R. A., & Brown, G. K. (1996). Beck Depression Inventory. San Antonio, TX: The Psychological Corporation.
- [Background] Belgrade, M., & Smith, S. (2013). Acupuncture and alternative treatments for painful diabetic neuropathy. Painful Diabetic Polyneuropathy, 83-93.
- [Background] Brown WJ, Dewey D, Bunnell BE, Boyd SJ, Wilkerson AK, Mitchell MA, Bruce SE. A Critical Review of Negative Affect and the Application of CBT for PTSD. Trauma Violence Abuse. 2018 Apr;19(2):176-194. doi: 10.1177/1524838016650188. Epub 2016 Jun 14. PMID 27301345
- [Background] Brown KW, Ryan RM. The benefits of being present: mindfulness and its role in psychological well-being. J Pers Soc Psychol. 2003 Apr;84(4):822-48. doi: 10.1037/0022-3514.84.4.822. PMID 12703651
- [Background] Brown, K. W., & Ryan, R. M. (2006). The Mindfulness Attention Awareness Scale (MAAS). Acceptance and Commitment Therapy. Measures Package, 82.
- [Background] Buysse DJ, Reynolds CF 3rd, Monk TH, Berman SR, Kupfer DJ. The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research. Psychiatry Res. 1989 May;28(2):193-213. doi: 10.1016/0165-1781(89)90047-4. PMID 2748771
- [Background] Chen LP, Murad MH, Paras ML, Colbenson KM, Sattler AL, Goranson EN, Elamin MB, Seime RJ, Shinozaki G, Prokop LJ, Zirakzadeh A. Sexual abuse and lifetime diagnosis of psychiatric disorders: systematic review and meta-analysis. Mayo Clin Proc. 2010 Jul;85(7):618-29. doi: 10.4065/mcp.2009.0583. Epub 2010 May 10. PMID 20458101
- [Background] Creswell JD. Mindfulness Interventions. Annu Rev Psychol. 2017 Jan 3;68:491-516. doi: 10.1146/annurev-psych-042716-051139. Epub 2016 Sep 28. PMID 27687118
- [Background] Derogatis, L. R., & Spencer, P. M. (1993). Brief Symptom Inventory: BSI. Upper Saddle River, NJ: Pearson.
- [Background] Diagnostic and Statistical Manual of Mental Disorders, (2013). American Psychiatric Publishing.
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Earley MD, Chesney MA, Frye J, Greene PA, Berman B, Kimbrough E. Mindfulness intervention for child abuse survivors: a 2.5-year follow-up. J Clin Psychol. 2014 Oct;70(10):933-41. doi: 10.1002/jclp.22102. Epub 2014 May 20. PMID 24844944
- [Background] Engel CC, Cordova EH, Benedek DM, Liu X, Gore KL, Goertz C, Freed MC, Crawford C, Jonas WB, Ursano RJ. Randomized effectiveness trial of a brief course of acupuncture for posttraumatic stress disorder. Med Care. 2014 Dec;52(12 Suppl 5):S57-64. doi: 10.1097/MLR.0000000000000237. PMID 25397825
- [Background] First, M. B., Spitzer, R. L., Gibbon, M., & Williams, J. B. W. (1996). Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-L Version 2.0). New York: Biometrics Research Department, New York State Psychiatric Institute.
- [Background] Flory JD, Yehuda R. Comorbidity between post-traumatic stress disorder and major depressive disorder: alternative explanations and treatment considerations. Dialogues Clin Neurosci. 2015 Jun;17(2):141-50. doi: 10.31887/DCNS.2015.17.2/jflory. PMID 26246789
- [Background] Foa, E.B., Hembree, E., & Rothbaum, B. (2007). Prolonged Exposiure Therapy for PTSD: Emotional Processing of Traumatic Experiences. Oxford University Press.
- [Background] Gallagher SM, Allen JJ, Hitt SK, Schnyer RN, Manber R. Six-month depression relapse rates among women treated with acupuncture. Complement Ther Med. 2001 Dec;9(4):216-8. doi: 10.1054/ctim.2001.0470. PMID 12184348
- [Background] Guy W. Clinical Global Impressions New Clinical Drug Evaluation Unit (ECDEU) Assessment Manual for Psychopharmacology - Revised. In: Department of Health E, and Welfare, Public Health Service, Alcohol, Drug Abuse, and Mental Health Administration, ed.; 1976:218-22.
- [Background] Hailes HP, Yu R, Danese A, Fazel S. Long-term outcomes of childhood sexual abuse: an umbrella review. Lancet Psychiatry. 2019 Oct;6(10):830-839. doi: 10.1016/S2215-0366(19)30286-X. Epub 2019 Sep 10. PMID 31519507
- [Background] Hirai K, Komura K, Tokoro A, Kuromaru T, Ohshima A, Ito T, Sumiyoshi Y, Hyodo I. Psychological and behavioral mechanisms influencing the use of complementary and alternative medicine (CAM) in cancer patients. Ann Oncol. 2008 Jan;19(1):49-55. doi: 10.1093/annonc/mdm494. Epub 2007 Oct 26. PMID 17965113
- [Background] Hollifield M. Acupuncture for posttraumatic stress disorder: conceptual, clinical, and biological data support further research. CNS Neurosci Ther. 2011 Dec;17(6):769-79. doi: 10.1111/j.1755-5949.2011.00241.x. Epub 2011 Feb 26. PMID 22070661
- [Background] Hollifield M, Sinclair-Lian N, Warner TD, Hammerschlag R. Acupuncture for posttraumatic stress disorder: a randomized controlled pilot trial. J Nerv Ment Dis. 2007 Jun;195(6):504-13. doi: 10.1097/NMD.0b013e31803044f8. PMID 17568299
- [Background] Kadel R. P., Kip K. E. (2012). A SAS Macro to Compute Effect Size (Cohen's) and its Confidence Interval from Raw Survey Data. Proceedings of the annual Southeastern SAS users Group Conference.
- [Background] Kar N. Cognitive behavioral therapy for the treatment of post-traumatic stress disorder: a review. Neuropsychiatr Dis Treat. 2011;7:167-81. doi: 10.2147/NDT.S10389. Epub 2011 Apr 4. PMID 21552319
- [Background] Kessler RC, Sonnega A, Bromet E, Hughes M, Nelson CB. Posttraumatic stress disorder in the National Comorbidity Survey. Arch Gen Psychiatry. 1995 Dec;52(12):1048-60. doi: 10.1001/archpsyc.1995.03950240066012. PMID 7492257
- [Background] Kessler RC, Chiu WT, Demler O, Merikangas KR, Walters EE. Prevalence, severity, and comorbidity of 12-month DSM-IV disorders in the National Comorbidity Survey Replication. Arch Gen Psychiatry. 2005 Jun;62(6):617-27. doi: 10.1001/archpsyc.62.6.617. PMID 15939839
- [Background] Kim YD, Heo I, Shin BC, Crawford C, Kang HW, Lim JH. Acupuncture for posttraumatic stress disorder: a systematic review of randomized controlled trials and prospective clinical trials. Evid Based Complement Alternat Med. 2013;2013:615857. doi: 10.1155/2013/615857. Epub 2013 Feb 6. PMID 23476697
- [Background] Kimbrough E, Magyari T, Langenberg P, Chesney M, Berman B. Mindfulness intervention for child abuse survivors. J Clin Psychol. 2010 Jan;66(1):17-33. doi: 10.1002/jclp.20624. PMID 19998425
- [Background] Lengacher CA, Johnson-Mallard V, Post-White J, Moscoso MS, Jacobsen PB, Klein TW, Widen RH, Fitzgerald SG, Shelton MM, Barta M, Goodman M, Cox CE, Kip KE. Randomized controlled trial of mindfulness-based stress reduction (MBSR) for survivors of breast cancer. Psychooncology. 2009 Dec;18(12):1261-72. doi: 10.1002/pon.1529. PMID 19235193
- [Background] Luterek JA, Harb GC, Heimberg RG, Marx BP. Interpersonal rejection sensitivity in childhood sexual abuse survivors: mediator of depressive symptoms and anger suppression. J Interpers Violence. 2004 Jan;19(1):90-107. doi: 10.1177/0886260503259052. PMID 14680531
- [Background] Meinert, C. L. & Tonascia S. Clinical trials: Design, conduct and analysis. Oxford: University Press.1986.
- [Background] Najavits LM. The problem of dropout from "gold standard" PTSD therapies. F1000Prime Rep. 2015 Apr 2;7:43. doi: 10.12703/P7-43. eCollection 2015. PMID 26097716
- [Background] Nixon RD, Nearmy DM. Treatment of comorbid posttraumatic stress disorder and major depressive disorder: a pilot study. J Trauma Stress. 2011 Aug;24(4):451-5. doi: 10.1002/jts.20654. Epub 2011 Jul 13. PMID 21755543
- [Background] National Comorbidity Survey (2005) NCS-R appendix tables: Table 1. Lifetime prevalence of DSM-IV/WMH-CIDI disorders by sex and cohort. Table 2. Twelve-month prevalence of DSM-IV/WMH-CIDI disorders by sex and cohort. Accessed at: http://www.hcp.med.harvard.edu/ncs/publications.php
- [Background] National Center for PTSD. (2012). Using the PTSD checklist (PCL). VA National Center for PTSD, July, 2012. Available online: http://sph.umd.edu/sites/default/files/files/PTSDChecklistScoring.pdf [Accessed August 1, 2016].
- [Background] Ostacher MJ, Cifu AS. Management of Posttraumatic Stress Disorder. JAMA. 2019 Jan 15;321(2):200-201. doi: 10.1001/jama.2018.19290. No abstract available. PMID 30556838
- [Background] Paivio SC, Laurent C. Empathy and emotion regulation: reprocessing memories of childhood abuse. J Clin Psychol. 2001 Feb;57(2):213-26. doi: 10.1002/1097-4679(200102)57:23.0.co;2-b. PMID 11180148
- [Background] Resick, P.A., Monson, C.M., & Chard, K.M. (2016). Cognitive Processing Therapy for PTSD: A Comprehensive Manual. Guildford Press.
- [Background] Rothman, K., & Greenland, S. (1998). Modern epidemiology. Philadelphia, PA: Lippincott-Raven.
- [Background] Shalev A, Liberzon I, Marmar C. Post-Traumatic Stress Disorder. N Engl J Med. 2017 Jun 22;376(25):2459-2469. doi: 10.1056/NEJMra1612499. No abstract available. PMID 28636846
- [Background] Sniezek DP, Siddiqui IJ. Acupuncture for Treating Anxiety and Depression in Women: A Clinical Systematic Review. Med Acupunct. 2013 Jun;25(3):164-172. doi: 10.1089/acu.2012.0900. PMID 24761171
- [Background] Watts BV, Schnurr PP, Mayo L, Young-Xu Y, Weeks WB, Friedman MJ. Meta-analysis of the efficacy of treatments for posttraumatic stress disorder. J Clin Psychiatry. 2013 Jun;74(6):e541-50. doi: 10.4088/JCP.12r08225. PMID 23842024
- [Background] Weathers FW, Keane TM, Davidson JR. Clinician-administered PTSD scale: a review of the first ten years of research. Depress Anxiety. 2001;13(3):132-56. doi: 10.1002/da.1029. PMID 11387733
- [Background] Whiting M, Leavey G, Scammell A, Au S, King M. Using acupuncture to treat depression: a feasibility study. Complement Ther Med. 2008 Apr;16(2):87-91. doi: 10.1016/j.ctim.2007.07.005. Epub 2007 Sep 29. PMID 18514910
- [Background] Wood AM, White IR, Thompson SG. Are missing outcome data adequately handled? A review of published randomized controlled trials in major medical journals. Clin Trials. 2004;1(4):368-76. doi: 10.1191/1740774504cn032oa. PMID 16279275
- [Background] Yehuda R. (2001). Immune neuroanatomic neuroendocrine gender differences in PTSD. Program and abstracts of the 154th Annual Meeting of the American Psychiatric Association; May 5-10, 2001; New Orleans, Louisiana. Symposium 12A.